CLINICAL TRIAL: NCT04330157
Title: The Influence of Systemic Inflammation on the Analgesic Effect of Tramadol After Major Abdominal Surgery
Brief Title: Inflammation and Postoperative Tramadol Analgesia
Status: Completed | Type: Observational
Sponsor: Osijek University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: OsijekUH-6
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Results first posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: General Surgery
Keywords: Postoperative analgesia; tramadol; intensive care unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CRP, PCT. leukocyte count, lactate, arterial blood gas
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients will be admitted in the intensive care unit after major abdominal surgery. All patients will receive 100 mg of tramadol intravenously every 6 hours. Pain will be assessed before and half an hour after tramadol administration by verbal Numeric Rating Scale.

DETAILED DESCRIPTION:
To all patients included in the study from the blood sample taken prior to the operation the leukocytes counts, c-reactive protein (CRP), procalcitonin (PCT) and lactate level will be performed, as well as arterial blood gas analysis.

After admission to the intensive care unit, all patients will receive 100 mg of tramadol intravenously every 6 hours. Pain will be assessed before and half an hour after tramadol administration by verbal Numeric Rating Scale (NRS). Pain score will be compared between patients with and without systemic inflammation. Systemic inflammation is defined as fulfilling at least two of the following major criteria: fever > 38 oC or hypothermia < 36 oC, tachycardia > 90 beats/minute, pCO2 in arterial blood < 4.3 kPa and leukocytes > 12.000/mm3 or < 4.000/mm3. Also, preoperative values of CRP > 50 mg/L and PCT > 0.5 ng/ml was also considered systemic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* elective and emergency open abdominal surgery
* ICU admission

Exclusion Criteria:

* tramadol allergy
* surgery performed laparoscopically
* age younger of 18 years and older the 90 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included patients admitted in the intensive care unit after major abdominal surgery performed with open laparotomy.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nenad Nešković, Principal Investigator — Anesthesiologyst
Locations (1):
- University hospital centre Osijek, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barakat A. Revisiting Tramadol: A Multi-Modal Agent for Pain Management. CNS Drugs. 2019 May;33(5):481-501. doi: 10.1007/s40263-019-00623-5. PMID 31004280
- [Background] He ZX, Chen XW, Zhou ZW, Zhou SF. Impact of physiological, pathological and environmental factors on the expression and activity of human cytochrome P450 2D6 and implications in precision medicine. Drug Metab Rev. 2015;47(4):470-519. doi: 10.3109/03602532.2015.1101131. Epub 2015 Nov 16. PMID 26574146
- [Background] Gerbershagen HJ, Rothaug J, Kalkman CJ, Meissner W. Determination of moderate-to-severe postoperative pain on the numeric rating scale: a cut-off point analysis applying four different methods. Br J Anaesth. 2011 Oct;107(4):619-26. doi: 10.1093/bja/aer195. Epub 2011 Jun 30. PMID 21724620
- [Background] Mallick P, Taneja G, Moorthy B, Ghose R. Regulation of drug-metabolizing enzymes in infectious and inflammatory disease: implications for biologics-small molecule drug interactions. Expert Opin Drug Metab Toxicol. 2017 Jun;13(6):605-616. doi: 10.1080/17425255.2017.1292251. Epub 2017 Feb 22. PMID 28537216

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Included in the Study: The study included patients admitted to the ICU after major abdominal surgeries.
Period: Overall Study
Arm/Group | Patients Included in the Study
Started | 50
Completed | 43
Not Completed | 7
Not completed — Protocol Violation | 4
Not completed — Not extubated within 24 h postoperatively | 3

BASELINE CHARACTERISTICS:
Groups:
- Demographic Characteristics of the Patients: Demographic characteristics of the patients included and type of surgical procedures
Arm/Group | Demographic Characteristics of the Patients
Number analyzed (Participants) | 43
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 67 [59 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 43
  More than one race | 0
  Unknown or Not Reported | 0
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 26.1 [22.8 to 28]
Smoking status [Count of Participants; unit: Participants]
  Yes | 18
  No | 25
ASA status [Count of Participants; unit: Participants] — ASA I: A normal healthy patient; ASA II: A patient with severe systemic disease; ASA III: A patient with severe systemic disease; ASA IV: A patient with severe systemic disease that is a constant threat to life.
  Participants
    II | 10
    III | 26
    IV | 7
Surgical procedure [Count of Participants; unit: Participants]
  Colorectal | 24
  Gastric | 6
  Small intestine | 2
  Liver | 5
  Pancreas | 3
  Multiple resection | 3

OUTCOME MEASURES:

1. Primary Outcome: Analgesic Affect of Tramadol After Major Abdominal Surgery
Description: Pain will be assessed before and half an hour after tramadol administration in awake patients by verbal Numeric Rating Scale. This scale has values from 0 to 10, where 0 means no pain and 10 means maximum pain.
Time Frame: NRS was assessed before and 30 minutes after each tramadol dose during first 24 postoperative hours
Population: NRS score was determinated only in awake patients
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Groups:
- NRS Score Before Tramadol Application: Before administration of tramadol to all patients who were extubated an NRS score was determined
- NRS Score After Tramadol Application: 30 minutes after administration of tramadol to all patients who were extubated an NRS score was determined
Arm/Group | NRS Score Before Tramadol Application | NRS Score After Tramadol Application
Number analyzed (Participants) | 43 | 43
Score on a scale
  1st assessment: number analyzed (Participants) | 8 | 12
  1st assessment | 7 [3.5 to 9.5] | 5 [4.25 to 6]
  2nd assessment: number analyzed (Participants) | 37 | 37
  2nd assessment | 5 [3 to 6.5] | 3 [1 to 5]
  3rd assessment: number analyzed (Participants) | 41 | 41
  3rd assessment | 4 [2.5 to 5] | 2 [1 to 3]
  4th assessment: number analyzed (Participants) | 42 | 41
  4th assessment | 4 [2 to 5] | 2 [1 to 4]
  5th assessment | 3 [2 to 5] | 2 [0 to 3]

2. Primary Outcome: Examine Differences in the Analgesic Effect of Tramadol Between Patients With and Without Postoperative Systemic Inflammation
Description: Differences in Numeric Rating Scale (NRS) in Patients with and without Systemic Inflammation. This scale has values from 0 to 10, where 0 means no pain and 10 means maximum pain.
Time Frame: NRS was assessed before and 30 minutes after each dose of tramadol in a first 24 postoperative hour
Population: NRS was assessed only in awake patients
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- NRS Before Tramadol - no Systemic Inflammation: NRS score in a patient who did not meet the criteria for systemic inflammation, before tramadol administration
- NRS After Tramadol - no Systemic Inflammation: NRS score in a patient who did not meet the criteria for systemic inflammation, after tramadol administration
- NRS Before Tramadol - With Systemic Inflammation: NRS score in a patient who meet the criteria for systemic inflammation, before tramadol administration
- NRS After Tramadol - With Systemic Inflammation: NRS score in a patient who meet the criteria for systemic inflammation, after tramadol administration
Arm/Group | NRS Before Tramadol - no Systemic Inflammation | NRS After Tramadol - no Systemic Inflammation | NRS Before Tramadol - With Systemic Inflammation | NRS After Tramadol - With Systemic Inflammation
Number analyzed (Participants) | 28 | 28 | 15 | 15
score on a scale
  1st assessment: number analyzed (Participants) | 7 | 9 | 1 | 3
  1st assessment | 7 [3 to 10] | 5 [3.5 to 5] | 7 [7 to 7] | 7 [6 to 7]
  2nd assessment: number analyzed (Participants) | 26 | 26 | 11 | 11
  2nd assessment | 5.5 [3.57 to 7.25] | 3 [1 to 4.25] | 4 [3 to 5] | 2 [1 to 5]
  3rd assessment: number analyzed (Participants) | 28 | 28 | 13 | 13
  3rd assessment | 4 [3 to 5] | 2 [1.25 to 3] | 3 [2 to 5] | 2 [0.5 to 4]
  4th assessment: number analyzed (Participants) | 28 | 28 | 14 | 13
  4th assessment | 4 [2 to 5] | 2.5 [1 to 4] | 3 [2 to 7.25] | 2 [1 to 3.5]
  5th assessment | 3 [2 to 5.75] | 2 [0.25 to 3.57] | 3 [2 to 5] | 2 [0 to 3]

ADVERSE EVENTS:
Time Frame: 24 hours
Groups:
- Adverse Effect: Adverse effect of tramadol
Arm/Group | Adverse Effect
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 16/43
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Effect (N=43)
Postoperative nausea and/or vomiting (Gastrointestinal disorders) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/57/NCT04330157/Prot_SAP_000.pdf